CLINICAL TRIAL: NCT06002321
Title: Right Ventricular Dysfunction in Chronic Heart Failure: Clinical Laboratory and Echocardiographic Characteristics
Brief Title: Right Ventricular Dysfunction in Chronic Heart Failure
Acronym: RIVED-CHF
Status: Not yet recruiting | Type: Observational
Sponsor: University of Siena (Other)
Collaborators: Italian Society of Cardiology (Other)
Responsible Party: Principal Investigator, Alberto Palazzuoli MD PhD, Professor, University of Siena
Other Study IDs: RIVED - CHF
Record Dates: First submitted 2023-07-21; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Chronic Heart Failure; Right Ventricular Dysfunction; Right Heart Failure
MeSH Terms: conditions — Ventricular Dysfunction, Right; Heart Failure | interventions — Echocardiography; Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HFpEF: The HFpEF group includes patients with signs and/or symptoms of heart failure and LVEF > 50% and objective evidence of structural and/or functional cardiac abnormalities consistent with the presence of LV diastolic dysfunction/raised LV filling pressures, including raised natriuretic peptides.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Laboratory Test
- HFmrEF: The HFmrEF group includes patients with signs and/or symptoms of heart failure and LVEF 41-49%.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Laboratory Test
- HFrEF: The HFrEF group includes patients with signs and/or symptoms of heart failure and LVEF < 40%.
  Interventions: Diagnostic Test: Echocardiography; Diagnostic Test: Laboratory Test

INTERVENTIONS:
Diagnostic Test: Echocardiography — Patients will undergo echocardiographic examination. The ejection fraction will be calculated using Simpson's method. The E/e' ratio will be measured using the Doppler method. E/e' > 13 will be considered an expression of the increase in LVFP. TAPSE will be measured together with the peak tricuspid regurgitation velocity (TVR). Pulmonary arterial hypertension will be defined as TVR > 2.8 m/s. Estimation of right atrial pressure (eRAP) will be obtained based on the diameter and inspiratory collapsibility of the inferior vena cava.
Diagnostic Test: Laboratory Test — BNP, NT-proBNP and renal function.

SUMMARY:
The goal of this multi center observational prospective study is to analyze the concordance between the signs and symptoms of RHF and echocardiographic features of RVD in patient with heart failure. The main questions it aims to answer are:

1. to assess the incidence of RVH and RVD in each HF subtypes.
2. to evaluate prognostic impact ( in terms of cardiovascular mortality and HF hospitalization) of different RVD patterns during a mean followup period of 3 years
3. To investigate the incidence of different RV maladaptation ( isolated RV dilatation, isolated Pulmonary hypertension, combined pattern) in each HF groups and the related outcome.

Participants will follow by direct check up visit and/or virtual visits every 6 months for a mean follow-up period of 3 years.

DETAILED DESCRIPTION:
Right ventricular dysfunction (RVD) and pulmonary hypertension (PH) have been recognized as two important prognostic features in patients with left side heart failure (HF). Nevertheless literature does not distinguish between right heart failure (RHF) and RVD, and the two terms are indifferently employed to describe PH and impaired RV performance. This is a multicenter observational prospective study endorsed by the Italian Society of Cardiology that would analyse the concordance between the signs and symptoms of RHF and echocardiographic features of RVD. Therefore the right ventricle (RV) adaptation across different left ventricular ejection fraction (LVEF) values, is poorly investigated. According to the recent heart failure (HF) guidelines classified patients based on LVEF in HF with preserved ( HFpEF) mild reduced (HFmEF) and reduced LVEF ( HFrEF), the investigators would assess by seral clinical laboratory and detailed echocardiographic study all patients affected by chronic HF regardless LVEF threshold in stable condition and will follow by direct check up visit and/or virtual visits every 6 months for a mean follow-up period of 3 years. All clinical laboratory and echocardiographic data will be recorded in a web platform system accessible for all center included in the study The main aims of the study are; 1- to assess the incidence of RVH and RVD in each HF subtypes. 2- to evaluate prognostic impact ( in terms of cardiovascular mortality and HF hospitalization) of different RVD patterns during a mean followup period of 3 years 3- To investigate the incidence of different RV maladaptation ( isolated RV dilatation, isolated Pulmonary hypertension, combined pattern) in each HF groups and the related outcome. The investigators expect to find different RVD degree and severity according to the type of left HF and its severity. Additionally, by a serial multiparametric analysis of RV, it would be possible to establish the stage and type of RVD and consequent concordance with signs of RHF.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a diagnosis of chronic heart failure made according to the recommendations of the ESC guidelines through the simultaneous presence of signs and symptoms of disease associated with BNP and NT proBNP levels > 100 and 300 pg/ml respectively which are associated with a modest increase PAPS > 30 mmHg with or without right ventricular dilatation.

Exclusion Criteria:

* Patients with dyspnea of non-cardiogenic origin, related to systemic respiratory diseases, pulmonary embolism, patients with primary pulmonary hypertension will be excluded.
* Patients with heart failure linked to primary valvular pathologies or infiltrative pathologies, secondary and on a genetic basis, patients diagnosed with acute heart failure in non-optimized therapy for at least 3 months will also be excluded. - Patients with systemic inflammatory neoplastic diseases, advanced liver and kidney diseases awaiting transplantation will be excluded.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with chronic heart failure will be consecutively enrolled prospectively in different cities. The diagnosis will be made on the basis of the signs and symptoms of the disease associated with BNP and NT-proBNP levels. Patients will be classified according to the type of cardiac structure and remodeling defect and ejection fraction.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Different patterns of RVD in chronic heart failure. | 6 months.
  The different patterns of RVD will be evaluated with echocardiographic measurements. Right ventricular function will be assessed by the following echocardiographic parameters: tricuspid annular plane excursion (TAPSE) and right ventricular fractional area change (RVFAC).
Analyze the incidence and prevalence of RVD and RHF. | 6 months.
  To analyze the incidence and prevalence of RVD and RHF according to left ventricular ejection fraction (HFrEF, HFmrEF, HFpEF).
Compare the clinical signs of right heart failure with the echocardiographic signs of RVD. | 6 months.
  Compare clinical signs of right heart failure with echocardiographic parameters of right ventricular dysfunction in order to verify agreement and identify a precise relationship between RHF and RVD.

SECONDARY OUTCOMES:
Define the incidence of RVD. | 6 months.
  To define the incidence of RVD through a multiparametric echocardiographic analysis including all the echocardiographic parameters of right ventricular function in order to identify a precise score based on the simultaneous dysfunction of several parameters.
Investigate a correlation between the different parameters. | 6 months.
  Investigate a correlation between echo parameters, clinical signs and laboratory data.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Palazzuoli, MD, Study Director — Unità di Malattie Cardiovascolari, Dipartimento Cardio-Toraco-Vascolare AOUS, Siena
Locations (14):
- Italy (14):
  - Centro Cardiologico Monzino, Milan, Milano
  - Department of Medicine, Surgery and Dentistry, Università di Salerno, Fisciano, Salerno
  - SC Universitaria di Cardiologia - UTIC Policlinico Riuniti Foggia, Foggia
  - Department of Clinical and Experimental Medicine, Operativee Unit of Cardiology, University of Messina, Messina
  - Ospedale Sant'Agostino Milano, Milan
  - Department of Translational Medical Sciences, CIRCET, Napoli
  - Department of Translational Medical Sciences, Federico II University, CIRCET, Napoli
  - Heart Failure Unit, Department of Cardiology, AORN dei Colli-Monaldi, Napoli
  - Fondazione IRCCS Policlinico San Matteo - Pavia UOC Cardiologia 1, Pavia
  - S. Maria della Misericordia Hospital, Perugia
  - SC Cardiologia, Azienda Ospedaliera Ospedale San Carlo Potenza, Potenza
  - Cardiology, Department of Clinica, Internal, Anesthesiology and Cardiovascular Scienses, Sapienza., Roma
  - Cardiology, Department of Clinica, Internal, Anesthesiology and Cardiovascular Scienses., Roma
  - Unità di Malattie Cardiovascolari, Dipartimento Cardio-Toraco-Vascolare AOUS, Università degli Studi, Siena., Siena

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Furey SA 3rd, Zieske HA, Levy MN. The essential function of the right ventricle. Am Heart J. 1984 Feb;107(2):404-10. doi: 10.1016/0002-8703(84)90402-2. No abstract available. PMID 6695680
- [Background] Poels EM, da Costa Martins PA, van Empel VP. Adaptive capacity of the right ventricle: why does it fail? Am J Physiol Heart Circ Physiol. 2015 Apr 15;308(8):H803-13. doi: 10.1152/ajpheart.00573.2014. Epub 2015 Feb 13. PMID 25681425
- [Background] Haddad F, Doyle R, Murphy DJ, Hunt SA. Right ventricular function in cardiovascular disease, part II: pathophysiology, clinical importance, and management of right ventricular failure. Circulation. 2008 Apr 1;117(13):1717-31. doi: 10.1161/CIRCULATIONAHA.107.653584. No abstract available. PMID 18378625
- [Background] Meyer P, Filippatos GS, Ahmed MI, Iskandrian AE, Bittner V, Perry GJ, White M, Aban IB, Mujib M, Dell'Italia LJ, Ahmed A. Effects of right ventricular ejection fraction on outcomes in chronic systolic heart failure. Circulation. 2010 Jan 19;121(2):252-8. doi: 10.1161/CIRCULATIONAHA.109.887570. Epub 2010 Jan 4. PMID 20048206
- [Background] Voelkel NF, Gomez-Arroyo J, Abbate A, Bogaard HJ. Mechanisms of right heart failure-A work in progress and a plea for failure prevention. Pulm Circ. 2013 Jan;3(1):137-43. doi: 10.4103/2045-8932.109957. No abstract available. PMID 23662190
- [Background] Markel TA, Wairiuko GM, Lahm T, Crisostomo PR, Wang M, Herring CM, Meldrum DR. The right heart and its distinct mechanisms of development, function, and failure. J Surg Res. 2008 May 15;146(2):304-13. doi: 10.1016/j.jss.2007.04.003. Epub 2007 Nov 26. PMID 18036544
- [Background] Ghio S, Acquaro M, Agostoni P, Ambrosio G, Carluccio E, Castiglione V, Colombo D, D'Alto M, Delle Grottaglie S, Dini FL, Emdin M, Fortunato M, Guaricci AI, Jacoangeli F, Marra AM, Paolillo S, Papa S, Scajola LV, Correale M, Palazzuoli A. Right heart failure in left heart disease: imaging, functional, and biochemical aspects of right ventricular dysfunction. Heart Fail Rev. 2023 Jul;28(4):1009-1022. doi: 10.1007/s10741-022-10276-0. Epub 2022 Nov 16. PMID 36385328
- [Background] de Groote P, Millaire A, Foucher-Hossein C, Nugue O, Marchandise X, Ducloux G, Lablanche JM. Right ventricular ejection fraction is an independent predictor of survival in patients with moderate heart failure. J Am Coll Cardiol. 1998 Oct;32(4):948-54. doi: 10.1016/s0735-1097(98)00337-4. PMID 9768716
- [Background] Gorter TM, van Veldhuisen DJ, Bauersachs J, Borlaug BA, Celutkiene J, Coats AJS, Crespo-Leiro MG, Guazzi M, Harjola VP, Heymans S, Hill L, Lainscak M, Lam CSP, Lund LH, Lyon AR, Mebazaa A, Mueller C, Paulus WJ, Pieske B, Piepoli MF, Ruschitzka F, Rutten FH, Seferovic PM, Solomon SD, Shah SJ, Triposkiadis F, Wachter R, Tschope C, de Boer RA. Right heart dysfunction and failure in heart failure with preserved ejection fraction: mechanisms and management. Position statement on behalf of the Heart Failure Association of the European Society of Cardiology. Eur J Heart Fail. 2018 Jan;20(1):16-37. doi: 10.1002/ejhf.1029. Epub 2017 Oct 16. PMID 29044932
- [Background] Nagueh SF, Bhatt R, Vivo RP, Krim SR, Sarvari SI, Russell K, Edvardsen T, Smiseth OA, Estep JD. Echocardiographic evaluation of hemodynamics in patients with decompensated systolic heart failure. Circ Cardiovasc Imaging. 2011 May;4(3):220-7. doi: 10.1161/CIRCIMAGING.111.963496. Epub 2011 Mar 11. PMID 21398512
- [Background] Sanz J, Sanchez-Quintana D, Bossone E, Bogaard HJ, Naeije R. Anatomy, Function, and Dysfunction of the Right Ventricle: JACC State-of-the-Art Review. J Am Coll Cardiol. 2019 Apr 2;73(12):1463-1482. doi: 10.1016/j.jacc.2018.12.076. PMID 30922478
- [Background] Drazner MH, Hamilton MA, Fonarow G, Creaser J, Flavell C, Stevenson LW. Relationship between right and left-sided filling pressures in 1000 patients with advanced heart failure. J Heart Lung Transplant. 1999 Nov;18(11):1126-32. doi: 10.1016/s1053-2498(99)00070-4. PMID 10598737
- [Background] Melenovsky V, Hwang SJ, Lin G, Redfield MM, Borlaug BA. Right heart dysfunction in heart failure with preserved ejection fraction. Eur Heart J. 2014 Dec 21;35(48):3452-62. doi: 10.1093/eurheartj/ehu193. Epub 2014 May 29. PMID 24875795
- [Background] Bosch L, Lam CSP, Gong L, Chan SP, Sim D, Yeo D, Jaufeerally F, Leong KTG, Ong HY, Ng TP, Richards AM, Arslan F, Ling LH. Right ventricular dysfunction in left-sided heart failure with preserved versus reduced ejection fraction. Eur J Heart Fail. 2017 Dec;19(12):1664-1671. doi: 10.1002/ejhf.873. Epub 2017 Jun 8. PMID 28597497
- [Background] Gorter TM, Hoendermis ES, van Veldhuisen DJ, Voors AA, Lam CS, Geelhoed B, Willems TP, van Melle JP. Right ventricular dysfunction in heart failure with preserved ejection fraction: a systematic review and meta-analysis. Eur J Heart Fail. 2016 Dec;18(12):1472-1487. doi: 10.1002/ejhf.630. Epub 2016 Sep 20. PMID 27650220
- [Background] Guazzi M, Borlaug BA. Pulmonary hypertension due to left heart disease. Circulation. 2012 Aug 21;126(8):975-90. doi: 10.1161/CIRCULATIONAHA.111.085761. No abstract available. PMID 22908015
- [Background] Konstam MA, Kiernan MS, Bernstein D, Bozkurt B, Jacob M, Kapur NK, Kociol RD, Lewis EF, Mehra MR, Pagani FD, Raval AN, Ward C; American Heart Association Council on Clinical Cardiology; Council on Cardiovascular Disease in the Young; and Council on Cardiovascular Surgery and Anesthesia. Evaluation and Management of Right-Sided Heart Failure: A Scientific Statement From the American Heart Association. Circulation. 2018 May 15;137(20):e578-e622. doi: 10.1161/CIR.0000000000000560. Epub 2018 Apr 12. PMID 29650544
- [Background] Puwanant S, Priester TC, Mookadam F, Bruce CJ, Redfield MM, Chandrasekaran K. Right ventricular function in patients with preserved and reduced ejection fraction heart failure. Eur J Echocardiogr. 2009 Aug;10(6):733-7. doi: 10.1093/ejechocard/jep052. Epub 2009 May 13. PMID 19443468
- [Background] Barilli M, Tavera MC, Valente S, Palazzuoli A. Structural and Hemodynamic Changes of the Right Ventricle in PH-HFpEF. Int J Mol Sci. 2022 Apr 20;23(9):4554. doi: 10.3390/ijms23094554. PMID 35562945
- [Background] Dini FL, Pugliese NR, Ameri P, Attanasio U, Badagliacca R, Correale M, Mercurio V, Tocchetti CG, Agostoni P, Palazzuoli A; Heart Failure Study Group of the Italian Society of Cardiology. Right ventricular failure in left heart disease: from pathophysiology to clinical manifestations and prognosis. Heart Fail Rev. 2023 Jul;28(4):757-766. doi: 10.1007/s10741-022-10282-2. Epub 2022 Oct 26. PMID 36284079
- [Background] Schmeisser A, Rauwolf T, Groscheck T, Kropf S, Luani B, Tanev I, Hansen M, Meissler S, Steendijk P, Braun-Dullaeus RC. Pressure-volume loop validation of TAPSE/PASP for right ventricular arterial coupling in heart failure with pulmonary hypertension. Eur Heart J Cardiovasc Imaging. 2021 Jan 22;22(2):168-176. doi: 10.1093/ehjci/jeaa285. PMID 33167032
- [Background] Guazzi M, Bandera F, Pelissero G, Castelvecchio S, Menicanti L, Ghio S, Temporelli PL, Arena R. Tricuspid annular plane systolic excursion and pulmonary arterial systolic pressure relationship in heart failure: an index of right ventricular contractile function and prognosis. Am J Physiol Heart Circ Physiol. 2013 Nov 1;305(9):H1373-81. doi: 10.1152/ajpheart.00157.2013. Epub 2013 Aug 30. PMID 23997100
- [Background] Guazzi M, Dixon D, Labate V, Beussink-Nelson L, Bandera F, Cuttica MJ, Shah SJ. RV Contractile Function and its Coupling to Pulmonary Circulation in Heart Failure With Preserved Ejection Fraction: Stratification of Clinical Phenotypes and Outcomes. JACC Cardiovasc Imaging. 2017 Oct;10(10 Pt B):1211-1221. doi: 10.1016/j.jcmg.2016.12.024. Epub 2017 Apr 12. PMID 28412423
- [Background] Gheorghiade M, Follath F, Ponikowski P, Barsuk JH, Blair JE, Cleland JG, Dickstein K, Drazner MH, Fonarow GC, Jaarsma T, Jondeau G, Sendon JL, Mebazaa A, Metra M, Nieminen M, Pang PS, Seferovic P, Stevenson LW, van Veldhuisen DJ, Zannad F, Anker SD, Rhodes A, McMurray JJ, Filippatos G; European Society of Cardiology; European Society of Intensive Care Medicine. Assessing and grading congestion in acute heart failure: a scientific statement from the acute heart failure committee of the heart failure association of the European Society of Cardiology and endorsed by the European Society of Intensive Care Medicine. Eur J Heart Fail. 2010 May;12(5):423-33. doi: 10.1093/eurjhf/hfq045. Epub 2010 Mar 30. PMID 20354029
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Lang RM, Badano LP, Mor-Avi V, Afilalo J, Armstrong A, Ernande L, Flachskampf FA, Foster E, Goldstein SA, Kuznetsova T, Lancellotti P, Muraru D, Picard MH, Rietzschel ER, Rudski L, Spencer KT, Tsang W, Voigt JU. Recommendations for cardiac chamber quantification by echocardiography in adults: an update from the American Society of Echocardiography and the European Association of Cardiovascular Imaging. J Am Soc Echocardiogr. 2015 Jan;28(1):1-39.e14. doi: 10.1016/j.echo.2014.10.003. PMID 25559473
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859
- [Background] Harjola VP, Mebazaa A, Celutkiene J, Bettex D, Bueno H, Chioncel O, Crespo-Leiro MG, Falk V, Filippatos G, Gibbs S, Leite-Moreira A, Lassus J, Masip J, Mueller C, Mullens W, Naeije R, Nordegraaf AV, Parissis J, Riley JP, Ristic A, Rosano G, Rudiger A, Ruschitzka F, Seferovic P, Sztrymf B, Vieillard-Baron A, Yilmaz MB, Konstantinides S. Contemporary management of acute right ventricular failure: a statement from the Heart Failure Association and the Working Group on Pulmonary Circulation and Right Ventricular Function of the European Society of Cardiology. Eur J Heart Fail. 2016 Mar;18(3):226-41. doi: 10.1002/ejhf.478. PMID 26995592
- [Background] Drazner MH, Rame JE, Stevenson LW, Dries DL. Prognostic importance of elevated jugular venous pressure and a third heart sound in patients with heart failure. N Engl J Med. 2001 Aug 23;345(8):574-81. doi: 10.1056/NEJMoa010641. PMID 11529211
- [Background] Ghio S, Guazzi M, Scardovi AB, Klersy C, Clemenza F, Carluccio E, Temporelli PL, Rossi A, Faggiano P, Traversi E, Vriz O, Dini FL; all investigators. Different correlates but similar prognostic implications for right ventricular dysfunction in heart failure patients with reduced or preserved ejection fraction. Eur J Heart Fail. 2017 Jul;19(7):873-879. doi: 10.1002/ejhf.664. Epub 2016 Nov 17. PMID 27860029
- [Background] Guazzi M, Naeije R. Pulmonary Hypertension in Heart Failure: Pathophysiology, Pathobiology, and Emerging Clinical Perspectives. J Am Coll Cardiol. 2017 Apr 4;69(13):1718-1734. doi: 10.1016/j.jacc.2017.01.051. PMID 28359519
- [Derived] Palazzuoli A, Dini FL, Agostoni P, Cartocci A, Morrone F, Tricarico L, Correale M, Mercurio V, Nodari S, Severino P, Badagliacca R, Barilla F, Paolillo S, Filardi PP; Italian Heart Failure Study Group, Italian Society of Cardiology. Right ventricular dysfunction in chronic heart failure: clinical laboratory and echocardiographic characteristics. (the RIVED-CHF registry). J Cardiovasc Med (Hagerstown). 2024 Jun 1;25(6):457-465. doi: 10.2459/JCM.0000000000001623. Epub 2024 Apr 26. PMID 38652523